CLINICAL TRIAL: NCT04595916
Title: A Multicenter, Randomized, Single-blind, Active-controlled Trial of The Efficacy and Safety of Polyene Phosphatidylcholine in Patients With Acute Drug-induced Liver Injury
Brief Title: Efficacy and Safety of Polyene Phosphatidylcholine in Treatment of Patients With Acute Drug-induced Liver Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSK-28-201
Record Dates: First submitted 2020-10-14; First posted 2020-10-22 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Acute Drug Induced Liver Injury
Keywords: ADILI
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury | interventions — polyene phosphatidylcholine; 18alpha,20beta-hydroxy-11-oxo-norolean-12-en-3beta-yl-2-O-beta-D-glucopyranurosyl-alpha-D-glucopyranosiduronate magnesium tetrahydrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyene Phosphatidylcholine (Experimental)
  Interventions: Drug: Polyene phosphatidylcholine injection 930 mg QD
- Magnesium Isoglycyrrhizinate (Active Comparator)
  Interventions: Drug: Magnesium Isoglycyrrhizinate injection 200 mg QD

INTERVENTIONS:
Drug: Polyene phosphatidylcholine injection 930 mg QD — Polyene phosphatidylcholine injection 930mg, diluted with 5% glucose solution 250ml, once a day, at least 2 weeks but no more than 4 weeks.
  Arms: Polyene Phosphatidylcholine
Drug: Magnesium Isoglycyrrhizinate injection 200 mg QD — Magnesium isoglycyrrhizinate injection 200mg, diluted with 5% glucose solution 250ml, once a day, at least 2 weeks but no more than 4 weeks.
  Arms: Magnesium Isoglycyrrhizinate

SUMMARY:
The purpose of this study is to explore the efficacy and the safety of polyene phosphatidylcholine Injection in patients with acute drug-induced liver injury after 2-4 weeks of treatment.

DETAILED DESCRIPTION:
This study is a phase IV study in subjects with acute drug-induced liver injury. As designed, the study will include a screening period of up to 1 week, 2 to 4 weeks of treatment, and 1 week of safety follow-up. The eligible subjects will randomly be assigned to polyene phosphatidylcholine group or magnesium isoglycyrrhizinate group to receive single-blind treatment with a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 75 years, Male or female patients
* Alanine aminotransferase (ALT) ≥ 3 x upper limit of normal (ULN) and Total bilirubin (TBIL) ≤ 5 x upper limit of normal (ULN)
* The Roussel Uclaf Causality Assessment Method (RUCAM) score is more than or equal to 6 points. The patients with RUCAM score of 3-5 needs to be determined by all three investigators that the liver injury is likely to be caused by drugs
* The duration of the current liver injury does not exceed 6 months

Exclusion Criteria:

* Liver injury caused by other diseases, such as viral hepatitis, alcoholic and non-alcoholic fatty liver disease, or autoimmune liver disease
* Acute liver failure or liver function decompensation, such as hepatic encephalopathy, ascites, albumin is less than 35g / L, the international standardized ratio (INR) of thrombin is more than 1.5
* Anemia or thrombocytopenia, hemoglobin is below 80 g/L, platelet count below 50,000 platelets per microliter
* Serum creatinine is more than 1.5 times ULN
* Severe hypokalemia, severe hypernatremia
* Patients have severe uncontrolled hypertension
* Severe diseases of vital organs such as heart, lung, brain, kidney, and gastrointestinal tract
* Treatment with polyene phosphatidylcholine injection or magnesium isoglycyrrhizinate injection within 5 days before informed consent
* Allergy or intolerance to benzyl alcohol and study drugs
* With no ability to express their complaints, such as mental illness and severe neurosis patient
* Pregnant or breastfeeding women, fertile women or men are reluctant to use contraception to avoid pregnancy during the trial
* Participation in another trial within 3 months before informed consent
* Patients who are considered by the investigator as inappropriate for the trial for other reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-04-04 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Serum ALT normalization rate | After 2-4 weeks treatment
  The serum ALT normalization rate of treatment for 2-4 weeks

SECONDARY OUTCOMES:
The serum ALT normalization rate for 1, 2 and 3 weeks | After 1, 2 and 3 weeks treatment
Changes in serum ALT compared to the baseline for 1, 2, 3 and 4 weeks | After 1, 2, 3 and 4 weeks treatment
The ratio of subjects whose ALT declined more than 50% compared to the base line for 1, 2, 3 and 4 weeks | After 1, 2, 3 and 4 weeks treatment
The serum AST normalization rate for 1, 2, 3 and 4 weeks | After 1, 2, 3 and 4 weeks treatment
Changes in serum AST compared to the baseline for 1, 2, 3 and 4 weeks | After 1, 2, 3 and 4 weeks treatment
The serum TBIL normalization rate for 1, 2, 3 and 4 weeks | After 1, 2, 3 and 4 weeks treatment
Changes in serum TBIL compared to the baseline for 1, 2, 3 and 4 weeks | After 1, 2, 3 and 4 weeks treatment
Changes in serum ALP and GGT compared to the baseline for 1, 2, 3 and 4 weeks | After 1, 2, 3 and 4 weeks treatment
The Incidence of Treatment-Emergent Adverse Events over time | After 2 to 4 weeks of treatment and 1 week of safety follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Mao, M.D., Study Chair — RenJi Hospital
Locations (9):
- China (9):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Chest Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The Sixth People's Hospital of Zhengzhou, Zhengzhou, Henan
  - The Third Hospital of Zhenjiang Affiliated Jiangsu University, Zhenjiang, Jiangsu
  - Renji Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Tongji Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No